CLINICAL TRIAL: NCT00663286
Title: A Clinical Trial Evaluating the Safety and Efficacy of IDP-110 in Patients With Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dow Pharmaceutical Sciences (Industry)
Responsible Party: Barry M. Calvarese, MS / Vice President, Regulatory & Clinical Affairs, Dow Pharmaceutical Sciences, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DPSI-06-22-2006-017
Record Dates: First submitted 2008-04-15; First posted 2008-04-22 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin; Benzoyl Peroxide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: IDP-110
- 2 (Active Comparator)
  Interventions: Drug: Clindamycin
- 3 (Active Comparator)
  Interventions: Drug: Benzoyl peroxide
- 4 (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: IDP-110 — Topical application for 12 weeks
  Arms: 1
Drug: Clindamycin — Topical application for 12 weeks
  Arms: 2
Drug: Benzoyl peroxide — Topical application for 12 weeks
  Arms: 3
Drug: Vehicle — Topical application for 12 weeks
  Arms: 4

SUMMARY:
The purpose of this study is to assess the effectiveness of IDP-110 in treating patients with acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Presence of inflammatory and non-inflammatory lesions

Exclusion Criteria:

* Dermatological conditions of the face other than acne that could interfere with clinical evaluations
* Female subjects who are pregnant, nursing, planning a pregnancy, or become pregnant during the study

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1399 (Actual)
Dates: Start 2006-10; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in number of lesions | 12 weeks

SECONDARY OUTCOMES:
Change from baseline in global severity | 12 weeks

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - The Savin Center, PC, New Haven, Connecticut
  - Webster Dermatology, PA, Hockessin, Delaware
  - Skin Care Research, Inc., Boca Raton, Florida
  - Advanced Dermatology and Cosmetic Surgery, Clermont, Florida
  - North Florida Dermatology Associates, PA, Jacksonville, Florida
  - Advanced Dermatology and Cosmetic Surgery, Ormond Beach, Florida
  - Dermatology Research, Pinellas Park, Florida
  - Florida Dermatology Institute, West Palm Beach, Florida
  - Derm Center of Augusta, Augusta, Georgia
  - MedaPhase Inc., Newnan, Georgia
  - Gwinnett Clinical Research Center, Inc., Snellville, Georgia
  - DuPage Medical Group, Naperville, Illinois
  - Hudson Dermatology, Evansville, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Dermatology Specialists Research, Louisville, Kentucky
  - Michigan Center for Research Corp., Clinton Township, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Atlantic Dermatologic Associates, LLP, Brooklyn, New York
  - Office of Fran E. Cook-Bolden, MD, New York, New York
  - Helendale Dermatology and Medical Spa, Rochester, New York
  - Dermatology Associates of Rochester, Rochester, New York
  - DermResearch Center of New York, Stony Brook, New York
  - Central Sooner Research, Norman, Oklahoma
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - DermResearch, Inc., Austin, Texas
  - J & S Studies, Inc., Bryan, Texas
  - Thomas J. Stephens & Associates, Carrollton, Texas
  - Dallas Associated Dermatologists, Dallas, Texas
  - Education & Research Foundation, Lynchburg, Virginia
  - Virginia Clinical Research, Inc, Norfolk, Virginia
  - Madison Skin & Research, Inc., Madison, Wisconsin